CLINICAL TRIAL: NCT03831672
Title: Post Market Multi-Center Retrospective Research on Embolization of Intracranial Aneurysms With Pipeline Embolization Device in China (PLUS)
Brief Title: Post Market Multi-Center Retrospective Research on Embolization of Intracranial Aneurysms With Pipeline Embolization Device in China
Acronym: PLUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Neurosurgical Institute (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Henan Provincial People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Group of Brain Doctors (Unknown); Peking University International Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); Qilu Hospital of Shandong University (Other); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); RenJi Hospital (Other); Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Xinjian Yang, MD, Vice Chair of Department of Interventional Neuroradiology, Beijing Neurosurgical Institute
Other Study IDs: KY2018-098-01
Record Dates: First submitted 2019-01-28; First posted 2019-02-06 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Intracranial Aneurysm; Pipeline Embolization Device
Keywords: intracranial aneurysm; outcome; occlusion; Pipeline embolization device; endovascular treatment; flow diversion
MeSH Terms: conditions — Intracranial Aneurysm; Bites and Stings

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pipeline TM embolization device launched to China in 2014, and has been widely used to treat large width IA. Therefore, it is necessary to collect and analysis the clinical data to evaluate effectiveness and safety of its usage in Chinese population, and this may guide the clinical practice and meet the clinical needs better.

DETAILED DESCRIPTION:
Recent years, the rapid development of endovascular treatment, especially the introduction of blood flow diverter device, has led to a new step in the treatment of intracranial aneurysms. It is different from usual treatment concept, blood flow diverter device's innovation is guiding to its parent artery reconstruction by cutting into the blood flow velocity and flow rate to the IA, and, promote the forming of aneurysm cavity thrombosis and the Neointima growth of IA's neck, so that to achieve aneurysm treatment.

A number of multi-center clinical studies on Pipeline embolization devices (PED, Ev3 Company/Medtronic, USA) have been conducted in North America and Europe recently. Becske etc reported the result of one multi-center prospective clinical trial of North America (PUFS), the PED treats the complicated intracranial internal carotid artery aneurysm. At the time of 180 days, 1 year, 3 years follow-up, the complete occlusion rate were 73.6%, 86.8% and 93.4% respectively. O 'kelly etc. the study showed that the rate of subtotal occlusion over 1 year follow-up of PED treatment for complex intracranial aneurysms was 90%. Many studies have confirmed the effectiveness of PED in the treatment of complex intracranial aneurysms.

The main motivation to innovate the blood flow diverter device is to use it to treat some large or giant aneurysms, fusiform aneurysm which can't be treated well by ordinary interventional embolization methods. So, in the initial stage of the application, its indications are mainly focus on the large or giant aneurysms located in the internal carotid artery before the origin of the posterior communicating artery. In recent years, the blood flow diverter devices were already used to treat many kinds of IA in almost all parts of the brain, different sizes and with pathological changes, such as dissecting aneurysms and vesicular aneurysms.

Although there was already much clinical research evidence which proved the efficacy and safety of PipelineTM 's treatment to the aneurysm as the embolization device, but these data are all from the foreign population, there is still no published clinical evidence of large sample size clinical study of Chinese population. Pipeline has been widely used to treat large width IA. Therefore, it's meaningful to evaluate effectiveness and safety in Chinese population, and this may guide the clinical practice and meet the clinical needs better.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepting to participate the study
* Patients treated with Pipeline

Exclusion Criteria:

* Patients treated by parent vessel occlusion
* Patients treated by other stent
* Patients lacking 3-dimensional aneurysm images or the images not satisfied the simulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The trial is intended to conduct in 13 centers in China. The sample size of this study was calculated based on the embolization rate of aneurysm. According to the existing overseas research data, we assume that the one-year embolization rate of Pipeline treatment for aneurysms is about 70%. Under the condition that the allowable error is 10% and the inspection level is 0.05, 162 cases are needed in this study. Considering the heterogeneity of different centers, the further expanded sample size is 200 cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete aneurysm occlusion in 12 months | assessed at 12 months (plus or minus 3 months) after procedure
  Complete occlusion defined as no contrast in contact with the IA neck or with the wall of the IA sac
Occurrence of ipsilateral major stroke or neurovascular death in 12 months | assessed at 12 months (plus or minus 3 months) after procedure
  Including but not limited: Spontaneous rupture of the target aneurysm, Ipsilateral intracranial hemorrhage, Ischemic stroke, Symptomatic parent artery stenosis, Permanent cranial neuropathy

SECONDARY OUTCOMES:
Rate of Complete aneurysm occlusion in 6 months | assessed at 6 months (plus or minus 3 months) after procedure
  Complete occlusion defined as no contrast in contact with the IA neck or with the wall of the IA sac
Rate of Complete aneurysm occlusion in 24 months | assessed at 24 months (plus or minus 6 months) after procedure
  Complete occlusion defined as no contrast in contact with the IA neck or with the wall of the IA sac
Occurrence of ipsilateral major stroke or neurovascular death in 1 month | assessed at 1 month (plus or minus 0.5 month) after procedure
  Including but not limited: Spontaneous rupture of the target aneurysm, Ipsilateral intracranial hemorrhage, Ischemic stroke, Symptomatic parent artery stenosis, Permanent cranial neuropathy
Device-related neurologic adverse event in 12 months | assessed at 12 months (plus or minus 3 months) after procedure
  Including but not limited: Spontaneous rupture of the target aneurysm, Ipsilateral intracranial hemorrhage, Ischemic stroke, Symptomatic parent artery stenosis, Permanent cranial neuropathy
Occurrence of ipsilateral major stroke or neurovascular death in 24 months | assessed at 24 months (plus or minus 6 months) after procedure
  Including but not limited: Spontaneous rupture of the target aneurysm, Ipsilateral intracranial hemorrhage, Ischemic stroke, Symptomatic parent artery stenosis, Permanent cranial neuropathy

CONTACTS AND LOCATIONS:
Overall Officials: Xinjian Yang, MD, Principal Investigator — Beijing Neurosurgical Institute and Beijing Tiantan Hospital
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang Y, Zhang F, Turhon M, Huang J, Li M, Peng Q, Zheng Z, Liu J, Zhang Y, Liu J, Zhang H, Li T, Song D, Zhao Y, Aisha M, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Guan S. Treatment of Intracranial Vertebral Artery Dissecting Aneurysms Using Pipeline Embolization Devices : A Multicenter Cohort Study. Clin Neuroradiol. 2023 Dec;33(4):1105-1114. doi: 10.1007/s00062-023-01318-7. Epub 2023 Jun 28. PMID 37380901
- [Derived] Zhao Y, Lu J, Zhang H, Li T, Song D, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Liu J, Zhao Y. Pipeline Embolization Device for intracranial aneurysms presenting with mass effect: a large Chinese cohort. Stroke Vasc Neurol. 2024 Feb 27;9(1):50-58. doi: 10.1136/svn-2022-002213. PMID 37295810
- [Derived] Lu J, Zhao Y, Zhang H, Li T, Song D, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Liu J, Zhao Y. Learning curve in pipeline embolization device: results from the pipeline embolization device in China post-market multicentre registry study. Int J Surg. 2023 Aug 1;109(8):2159-2167. doi: 10.1097/JS9.0000000000000467. PMID 37158157
- [Derived] Zhang H, Li L, Zhang H, Liu J, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Luo B, Shao Q, Chang K, Zhang Q, He Y, Zhang P, Yang X, Li TX. Small and Medium-Sized Aneurysm Outcomes Following Intracranial Aneurysm Treatment Using the Pipeline Embolization Device: A Subgroup Analysis of the PLUS Registry. Front Neurol. 2022 May 31;13:881353. doi: 10.3389/fneur.2022.881353. eCollection 2022. PMID 35711259
- [Derived] Xu C, Wu P, Han J, Sun B, Wang C, Xu S, Luo B, Yang X, Mu Q, Shi H. Safety Evaluation and Flow Modification in the Anterior Cerebral Artery after Pipeline Embolization Device Deployment across the Internal Carotid Artery Terminus. Biomed Res Int. 2021 Aug 21;2021:6657595. doi: 10.1155/2021/6657595. eCollection 2021. PMID 34471639
- [Derived] Kang H, Luo B, Liu J, Wang A, Zhang H, Li T, Song D, Zhao Y, Guan S, Wang Y, Feng W, Wang Y, Shi H, Liu J, Yang X. A novel score for evaluating cerebral aneurysms treated with flow diversion: 4F-flow diversion predictive score. Ther Adv Neurol Disord. 2021 Aug 19;14:17562864211039336. doi: 10.1177/17562864211039336. eCollection 2021. PMID 34434256
- [Derived] Kang H, Zhou Y, Luo B, Lv N, Zhang H, Li T, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X, Liu J. Pipeline Embolization Device for Intracranial Aneurysms in a Large Chinese Cohort: Complication Risk Factor Analysis. Neurotherapeutics. 2021 Apr;18(2):1198-1206. doi: 10.1007/s13311-020-00990-8. Epub 2021 Jan 14. PMID 33447904
- [Derived] Luo B, Kang H, Zhang H, Li T, Liu J, Song D, Zhao Y, Guan S, Maimaitili A, Wang Y, Feng W, Wang Y, Wan J, Mao G, Shi H, Yang X. Pipeline Embolization device for intracranial aneurysms in a large Chinese cohort: factors related to aneurysm occlusion. Ther Adv Neurol Disord. 2020 Nov 2;13:1756286420967828. doi: 10.1177/1756286420967828. eCollection 2020. PMID 33224273